CLINICAL TRIAL: NCT04632602
Title: Awake Prone Position to Reduce Ventilation Inhomogeneity in COVID-19 Acute Respiratory Failure: a Randomized Cross Over Electrical Impedance Tomography Study
Brief Title: Awake Prone Position to Reduce Ventilation Inhomogeneity in COVID-19 Acute Respiratory Failure
Acronym: ProneSpontCov
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2020-17
Record Dates: First submitted 2020-11-16; First posted 2020-11-17 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Each patient will be his own control. The order of the experimental periods will be:
  1. arm A: prone position followed by dorsal decubitus
  2. arm B: dorsal decubitus followed by ventral decubitus A 30-minute wash-out period is set between the end of sequence 1 and the start of sequence 2.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients in prone position followed by dorsal decubitus (Other): patients will be randomized on the order of position, either supine then prone, either prone then supine. Each period will last at least 2 hours.
  Interventions: Other: physiological effects of awake prone position in COVID 19 patients
- dorsal decubitus followed by prone decubitus (Other): patients will be randomized on the order of position, either supine then prone, either prone then supine. Each period will last at least 2 hours.
  Interventions: Other: physiological effects of awake prone position in COVID 19 patients

INTERVENTIONS:
Other: physiological effects of awake prone position in COVID 19 patients — Study of physiological effects of awake prone position in COVID 19 patients on lung inhomogeneity assessed by Electrical Impedance Tomography (EIT), gas exchange and dyspnea score (Borg Scale).
  Measurements will be performed at baseline (on supine position), then patients will be randomized on the order of position, either supine then prone, either prone then supine. Each period will last at least 2 hours. EIT records will be performed during the last 30 minutes of each period, blood gas and dyspnea score at the end of each period.

SUMMARY:
Evaluation of awake prone position on ventilation inhomogeneity in COVID-19 associated respiratory failure.

DETAILED DESCRIPTION:
Awake prone position has been proposed as an additional treatment to alleviate hypoxemia during COVID-19 acute respiratory failure and potentially to avoid in some case tracheal intubation and invasive ventilation. Potential mechanism is improvement of ventilation: perfusion mismatch through redistribution of ventilation to the dorsal part of the lungs where perfusion is prominent. Electrical impedance tomography (EIT) is a non-invasive functional lung imaging of distribution of ventilation. Therefore, we aim to assess EIT on lung ventilation inhomogeneity during supine and prone position in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 Years (Adult, Older Adult)
* Confirmed COVID-19 (positive SARS-CoV-2 RT-PCR at nasopharyngeal swab)
* Acute respiratory failure with 100 < PaO2:FiO2< 300 mmhg
* Spontaneous ventilation with standard oxygen supply or high flow humidified oxygen
* Written informed consent of the patient

Exclusion Criteria:

* Contra-indication to prone position including pregnancy
* Presence of pacemaker
* Severe hypoxemia with PaO2/FiO2 < 100 mmHg
* Evidence of clinical signs of respiratory distress with high probability of intubation in the next two hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-11-29 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Global Inhomogeneity Index variations (expressed in percentage) between baseline, supine and prone position periods. | 2hours
  Electrical Impedance Tomography (EIT)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — ASSISTANCE PUBLIQUE HÔPITAUX DE MARSEILLE
Locations (1):
- Assistance Publique Höpitaux de Marseille, Marseille, France